CLINICAL TRIAL: NCT03543826
Title: Best Practice With Rocuronium, Neostigmine, Sugammadex, and Subjective Monitoring.
Brief Title: Best Practice Using Rocuronium and Reversal With Neostigmine or Sugammadex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Stephan Thilen, Associate Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003888
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Results first posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-05

CONDITIONS: Muscle Weakness
Keywords: neostigmine; sugammadex; rocuronium; neuromuscular blocking agents
MeSH Terms: conditions — Muscle Weakness | interventions — Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects undergoing orthopedic or abdominal surgery (Other): Subjects undergoing orthopedic or abdominal surgery requiring neuromuscular blockade. Subjects all receive the neuromuscular blockade drug Rocuronium based on study protocol. Depending on depth of block (subjectively assessed by TOF response), Neostigmine, Sugammadex, or no reversal drug is used to reverse block prior to extubation.
  Interventions: Combination Product: Protocol for rocuronium neuromuscular block

INTERVENTIONS:
Combination Product: Protocol for rocuronium neuromuscular block — The protocol includes specified appropriate rocuronium dosing and a valid pre-reversal assessment of the adductor pollicis response guides optimal neostigmine vs. sugammadex reversal.

SUMMARY:
This is an estimation study, prospectively evaluating the incidence of postoperative residual neuromuscular blockade (PRNB) when a best practice protocol is implemented for a cohort of abdominal surgery and orthopedic surgery patients. The protocol is developed within the constraint of subjective monitoring, quantitative monitoring is not used, and use of rocuronium for paralysis and either neostigmine or sugammadex for reversal. The primary outcome is the incidence of PRNB on arrival to the post-anesthesia care unit, defined as a train-of-four ration <0.9.

DETAILED DESCRIPTION:
This study estimates the incidence of postoperative residual neuromuscular block when rocuronium neuromuscular block is managed by protocol for qualitative monitoring and reversal with neostigmine or sugammadex. The study is an extension of the recently published study by Thilen and co-workers which evaluated a protocol which used neostigmine as the sole reversal agent (doi: 10.1016/j.bja.2018.03.029). It demonstrated that use of a protocol was associated with a reduced incidence of severe residual paralysis, defined as normalized train-of-four (TOF) ratio <0.7 at time of tracheal extubation. It was also associated with a highly significant reduction in PRNB as defined for several secondary outcomes, including non-normalized (i.e. raw) TOF-ratio <0.9 at time of arrival to the post-anesthesia care unit (PACU).

The current study does not include a control group, only an intervention group. The investigators hypothesize that PRNB can be prevented by adhering to a protocol which incorporates several current recommendations by experts. Importantly, the protocol preserves a role for neostigmine when the pre-reversal assessment indicates that spontaneous recovery has progressed to a so-called minimal block which is defined as the subjective absence of fade in the adductor pollicis TOF response. The investigators will study only abdominal surgery and orthopedic surgery patients. The primary outcome is incidence of PRNB, defined as TOF-ratio <0.9 on arrival to the PACU. The investigators plan to enroll 120 patients, and if no more than one patient has PRNB, the upper bound for the 95% confidence interval will be less than 5%.

ELIGIBILITY:
Inclusion Criteria: Adult 18 years old or older, Will undergo open or laparoscopic abdominal surgery or orthopedic surgery expected to last <6 hours at Harborview or Univ of Wash Med Ctr, Have American Society of Anesthesiologists physical status I-III, scheduled to have general anesthesia with at least 1 dose of nondepolarizing neuromuscular blocking drug for endotracheal intubation or intraoperative neuromuscular blockade.

-

Exclusion Criteria: Allergy to neuromuscular blocking drugs, patients with neuromuscular disease (myasthenia gravis or muscular dystrophy), pregnant or lactating women, non-English speaking.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan R Thilen, MD, MS, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thilen SR, Liang T, Kruse TN, Cain KC, Treggiari MM, Bhananker SM. Evaluation of a Protocol for the Management of Maintenance and Reversal of Rocuronium Block Using Neostigmine or Sugammadex. Anesth Analg. 2023 Jun 1;136(6):1143-1153. doi: 10.1213/ANE.0000000000006510. Epub 2023 May 19. PMID 37205804

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 201 subjects were consented to the study. However, 163 subjects completed the study and were included in the primary per-protocol analysis.
Period: Overall Study
Arm/Group | Subjects Undergoing Orthopedic or Abdominal Surgery
Started | 163
Completed | 163
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: We approached 201 patients who provided signed informed consent. A total of 163 patients completed the study and were included in the primary per-protocol analysis.
Arm/Group | Subjects Undergoing Orthopedic or Abdominal Surgery
Number analyzed (Participants) | 163
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 129
  >=65 years | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 13
  White | 135
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 163

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Postoperative Residual Neuromuscular Blockade at Time of Arrival to the Post-anesthesia Care Unit.
Description: Postoperative residual neuromuscular blockade is measured by a Train-of-four ratio <0.9 as measured by acceleromyography.
Time Frame: Within five minutes of arrival to the post-anesthesia care unit.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Undergoing Orthopedic or Abdominal Surgery
Number analyzed (Participants) | 163
Participants | 5

2. Secondary Outcome: Incidence of Postoperative Severe Residual Neuromuscular Blockade at Time of Arrival to the Post-anesthesia Care Unit.
Description: Postoperative severe residual neuromuscular blockade is measured by a Train-of-four ratio <0.7 as measured by acceleromyography.
Time Frame: Within five minutes of arrival to the post-anesthesia care unit.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Undergoing Orthopedic or Abdominal Surgery
Number analyzed (Participants) | 163
Participants | 2

3. Secondary Outcome: Incidence of Postoperative Residual Neuromuscular Blockade at Time of Tracheal Extubation.
Description: as for outcome 1
Time Frame: Within two minutes of time of extubation.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Undergoing Orthopedic or Abdominal Surgery
Number analyzed (Participants) | 161
Participants | 14

4. Secondary Outcome: Incidence of Postoperative Severe Residual Neuromuscular Blockade at Time of Tracheal Extubation
Description: as for outcome 2
Time Frame: Within two minutes of time of extubation.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Undergoing Orthopedic or Abdominal Surgery
Number analyzed (Participants) | 161
Participants | 1

ADVERSE EVENTS:
Time Frame: 1 day: Day of surgery through recovery in PACU.
Arm/Group | Subjects Undergoing Orthopedic or Abdominal Surgery
All-Cause Mortality (participants affected / at risk) | 0/163
Serious Adverse Events (participants affected / at risk) | 0/163
Other Adverse Events (participants affected / at risk) | 0/163

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT03543826/Prot_003.pdf
  • Statistical Analysis Plan (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT03543826/SAP_004.pdf
  • Informed Consent Form (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT03543826/ICF_005.pdf